CLINICAL TRIAL: NCT07178782
Title: Effect of Dual-task Training Program on Balance and Hand Functions in Unilateral Cerebral Palsy
Brief Title: Dual-Task Training for Balance and Hand Function in Unilateral CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, hanaa mohsen, assistant professor, Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hana 10
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Balance
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): selected rehabilitation program
  Interventions: Other: rehabilitation program
- intervention (Experimental): dual task exercises in the form of balance and hand functions
  Interventions: Other: Dual-Task Training Program

INTERVENTIONS:
Other: Dual-Task Training Program — the participant will receive dual task program in form of balance and hand function program
  Arms: intervention
Other: rehabilitation program — designed rehabilitation program
  Arms: control

SUMMARY:
This trial will evaluate the impact of a dual-task training program on children aged 6-8 years with unilateral cerebral palsy. Seventy participants will be randomized into dual-task and single-task groups, with the dual-task group performing balance exercises while engaging in fine motor tasks. It is expected that dual-task training will produce superior improvements in balance and hand function, offering a safe and effective alternative to traditional single-task methods.

ELIGIBILITY:
Inclusion Criteria:

* - Their age will range from 6 to 8 years.
* Mild degree of spasticity ranged from 1 to 1+ according to Modified Ashworth Scale
* Their motor function will be at level I and II according to Gross Motor Function Classification System GMFCS

Exclusion Criteria:

* - Botulinum toxin injections in the last 6 months.
* The presence of visual perceptual impairment.
* Surgical interference in upper, lower limbs and/or spine.
* Muscloskeletal problems or fixed deformities in the spine and/or upper or/and lower extremities.
* Seizures.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
HUMAC Balance | pre and post treatment 3 month
  humac balance
Bruininks-Oseretsky | pre and post treatment 3 month
  Fine motor Proficiency assessed by Bruininks-Oseretsky

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa M Abd-Elfattah, Principal Investigator — Associate professor
Locations (1):
- Badr Univesity in Cairo (BUC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No